CLINICAL TRIAL: NCT00451971
Title: Objective Study in Rheumatoid Arthritis
Acronym: OSRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HWA486_4020; NCT00251667 (obsolete NCT alias)
Record Dates: First submitted 2007-03-23; First posted 2007-03-26 (Estimated); Last update posted 2008-09-05 (Estimated); Status verified 2008-09

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Leflunomide

INTERVENTIONS:
Drug: LEFLUNOMIDE

SUMMARY:
Primary Objectives

1. To test the feasibility, in patients with active rheumatoid arthritis, of using an 'aggressive' treatment algorithm to bring a short term treatment objective (STO) within the normal or an arbitrarily defined 'desirable' range.
2. To determine whether patients with active rheumatoid arthritis randomly allocated to a particular STO show a reduced rate of Magnetic resonance imaging damage progression at two years compared to those randomly allocated to usual care.

Secondary Objectives

1. To establish the relationship between achieving a given STO or combination of STOs and damage progression.
2. To identify the characteristics of responders and non-responders with respect to STO achievement and predictors of greater and lesser degrees of damage progression.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid Arthritis as defined by the American College of Rhemuatology criteria and either
* Active disease: ≥6/28 swollen joints or
* Erythrocyte sedimantation or C-Reactive Protein > normal
* Disease duration ≤ 15 yrs
* Any therapy
* Females of child-bearing potential must be adequate contraception

Exclusion Criteria:

* Frailty, limiting co-morbidity
* Obesity limiting ability to have MRI
* Geographical difficulty preventing follow-up and visits
* Women at risk of becoming pregnant

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2002-03

PRIMARY OUTCOMES:
Long Term Objective (damage) is the MRI which will be undertaken at baseline, 12 months and 24 months.
The Short Term Objectives are: swollen joint count - target:(28) ≤ 2 joints
C-Reactive Protein - target: within the normal range (provided elevation is not due clinically to an intercurrent event)

SECONDARY OUTCOMES:
Safety: Full blood count and erythrocyte sedimentation, blood urea, electrolytes, creatinine and Liver function test

CONTACTS AND LOCATIONS:
Overall Officials: J Edmonds, Principal Investigator — Sanofi
Locations (1):
- Sanofi-Aventis, Sydney, Australia

REFERENCES:
- [Derived] Poh MQ, Lassere M, Bird P, Edmonds J. Reliability and longitudinal validity of computer-assisted methods for measuring joint damage progression in subjects with rheumatoid arthritis. J Rheumatol. 2013 Jan;40(1):23-9. doi: 10.3899/jrheum.120549. Epub 2012 Nov 1. PMID 23118111